CLINICAL TRIAL: NCT00584038
Title: Improving Adolescent Adherence to Hormonal Contraception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 06-060; R40MC06634
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Contraception
Keywords: contraceptive compliance; educational intervention; oral contraception
MeSH Terms: interventions — Ambulatory Care Facilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Standard Care (SC) (No Intervention): Participants receive usual contraceptive care administered by clinic provider.
- 2 Standard Care + Educational (SCE) (Other): Participants receive standard contraceptive care from clinic provider, followed by 45-minute educational intervention.
  Interventions: Behavioral: educational instruction in clinic
- 3 Standard Care + Educational + Phone Calls (SCEP) (Other): Participants receive standard contraceptive care from clinic provider, followed by phone calls weekly until onset of menses and monthly thereafter for six consecutive months.
  Interventions: Behavioral: educational instruction and phone follow-up

INTERVENTIONS:
Behavioral: educational instruction and phone follow-up — Educational instruction and phone follow-up.
  Arms: 3 Standard Care + Educational + Phone Calls (SCEP)
Behavioral: educational instruction in clinic — Educational instruction in clinic.
  Arms: 2 Standard Care + Educational (SCE)

SUMMARY:
The purpose of this study is to determine whether contraceptive compliance by young women can be improved through expanded counseling by a health educator at the initial clinic visit as compared with standard care.

ELIGIBILITY:
Inclusion criteria:

* Sexually active females 16 to 24 years of age who present to a University of Texas Medical Branch (UTMB) clinic and request to initiate oral contraception for birth control.

Exclusion criteria:

* Women who are currently pregnant or breastfeeding.
* Women who wish to become pregnant within the next 12 months.
* Women who have a medical contraindication to use of estrogen (e.g., thromboembolic disease, acute liver disease, breast cancer, genital cancer, or undiagnosed genital bleeding).
* Women wishing to initiate use of a contraceptive method that is not oral, such as transdermal (the patch) or injectable (DMPA) methods, or the vaginal ring.
* Current and previous users of oral contraceptives.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1155 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Measurement of contraceptive adherence | 12 months
Measurement of dual method use | 12 months
Measurement of pregnancy rates and sexually transmitted diseases (STDs) | 12 months

SECONDARY OUTCOMES:
Measurement of contraceptive side effects | 12 months
Measurement of satisfaction with method | 12 months
Measurement of sexual activity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abbey B. Berenson, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Berenson AB, Rahman M. A randomized controlled study of two educational interventions on adherence with oral contraceptives and condoms. Contraception. 2012 Dec;86(6):716-24. doi: 10.1016/j.contraception.2012.06.007. Epub 2012 Jul 25. PMID 22840278